CLINICAL TRIAL: NCT02661451
Title: Transcatheter Aortic Valve Replacement to UNload the Left Ventricle in Patients With ADvanced Heart Failure: A Randomized Trial (TAVR UNLOAD)
Brief Title: Transcatheter Aortic Valve Replacement to UNload the Left Ventricle in Patients With ADvanced Heart Failure (TAVR UNLOAD)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiovascular Research Foundation, New York (Other)
Collaborators: Cardialysis BV (Industry); Avania (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAVR Unload
Record Dates: First submitted 2016-01-15; First posted 2016-01-22 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Aortic Valve Stenosis
Keywords: Valve
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAVR (with SAPIEN 3 THV) and OHFT (Experimental): Transcatheter heart valve and Optimal Heart Failure Therapy
  Interventions: Device: SAPIEN 3 THV; Biological: Optimal Heart Failure Therapy
- OHFT (Active Comparator): Optimal Heart Failure Therapy
  Interventions: Biological: Optimal Heart Failure Therapy

INTERVENTIONS:
Device: SAPIEN 3 THV
  Arms: TAVR (with SAPIEN 3 THV) and OHFT
Biological: Optimal Heart Failure Therapy

SUMMARY:
The objective of this study is to determine the safety and efficacy of transcatheter aortic valve replacement (TAVR) via a transfemoral approach in HF patients with moderate AS as compared with OHFT.

ELIGIBILITY:
Inclusion Criteria

All candidates for this study must meet all of the following inclusion criteria:

1. Age ≥18 years
2. Heart Failure with NYHA class ≥ 2
3. Under appropriate and stable guideline-directed HF therapy for a minimum of 1 month prior to randomization.

   Note: Patients are expected to be on appropriate pharmacologic therapy and if indicated CRT for heart failure. (12, 13) Patients with aortic stenosis may not be able to tolerate maximal doses of heart failure medications and no specific guidelines exist for the medical treatment of heart failure in the setting of aortic stenosis. It is expected that the heart failure PI will review the medical therapy and confirm that it is appropriate for the patient's condition.
4. Moderate AS confirmed by the echo core lab. Moderate AS is defined as an aortic valve area (AVA) >1.0 cm2 and ≤1.5 cm2 on rest echo or if ≤1.0 cm2 at rest and low-flow AS is suspected when the an AVA > 1.0 cm2 with low dose dobutamine stress echo (DSE). Patients with AVA<1.0 cm2 but with an indexed AVA of >0.6 cm2/m2 on either rest or DSE are also eligible. Similarly, patients with AVA >1.5 cm2 but with indexed AVA<0.9 cm2/m2 on either rest of DSE are also eligible.

   Note: Typically such cases will demonstrate,

   • Mean trans-aortic gradient (MG) ≥ 20 mmHg and < 40 mmHg at rest and aortic valve area (AVA) > 1.0 cm2 and ≤1.5 cm2 (or AVA < 1.0 cm2 but indexed AVA > 0.6 cm2) at rest

   OR

   • Mean trans-aortic gradient (MG) ≥ 20 mmHg and < 40 mmHg and aortic valve area (AVA) ≤1.0 cm2 at rest AND MG < 40 mmHg and aortic valve area (AVA)

   •>1.0 cm2 (or AVA < 1.0 cm2 but indexed AVA > 0.6 cm2) with low dose dobutamine stress echo (DSE).

   In atypical cases (for example mean gradient is below 20 mmHg but valve area is consistent with moderate AS, the final eligibility determination in regards to diagnosis of moderate AS will be made by the echocardiographic core lab.
5. Left ventricular (LV) ejection fraction (EF) < 50% at rest
6. Anatomically suitable for transfemoral TAVR with the SAPIEN 3 or SAPIEN 3 Ultra THV
7. Able to provide independent informed consent (i.e., not requiring a legally authorized representative)

Exclusion Criteria

Candidates are excluded from the study if any of the following conditions are present:

1. LVEF < 20% or persistent need for intravenous inotropic support
2. Hospitalization for acute decompensated HF within 2 weeks prior to randomization
3. Cardiac resynchronization therapy (CRT) device implantation within 1 month prior to randomization
4. Coronary artery revascularization (PCI or CABG) within 1 month prior to randomization
5. In need and suitable for revascularization per heart team consensus
6. Severe aortic and/or mitral regurgitation
7. Congenital unicuspid or congenital bicuspid aortic valve
8. Concomitant non-aortic valvular disease with a formal indication for valve surgery per established guidelines (ESC/ACC/AHA)
9. Previous aortic valve replacement (mechanical or bioprosthetic)
10. Severe RV dysfunction
11. Previous stroke with permanent disability (modified Rankin score ≥ 2)
12. Severe lung disease as indicated by FEV1 <30% predicted or need for chronic daytime supplemental oxygen therapy
13. Severe chronic kidney disease: glomerular filtration rate (GFR) < 30 mL/min by MDRD or need for renal replacement therapy
14. Gastrointestinal (GI) bleeding within the past 3 months
15. Liver cirrhosis Child-Pugh C
16. Active systemic infection, including active endocarditis
17. Unwilling to accept blood transfusion
18. Evidence of intracardiac mass, thrombus or vegetation
19. Absence of minimum amount of aortic valve calcification necessary for TAVR with the SAPIEN 3 or SAPIEN 3 Ultra THV
20. Hypersensitivity or contraindication to clopidogrel, aspirin, or to oral anticoagulation if indicated (e.g. subject in atrial fibrillation)
21. Sensitivity to contrast media which cannot be adequately pre-medicated
22. Women of child-bearing potential
23. Clinical signs of dementia
24. Other medical, social, or psychological conditions that precludes appropriate consent and follow-up
25. Life expectancy < 2 years due to cancer or other non-cardiac chronic diseases
26. Unwillingness to undergo follow-up investigations
27. Currently participating in an investigational drug or another device trial that has not reached its primary endpoint (excluding registries)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
All-Cause Death | 12 months
  Hierarchical occurrence within efficacy assessment time interval (EATI) of:
Disabling Stroke | 12 months
  Hierarchical occurrence within efficacy assessment time interval (EATI) of:
Hospitalizations related to heart failure, symptomatic aortic valve disease or non-disabling stroke -or - Clinically significant worsening of heart failure (heart failure hospitalization equivalent). | 12 months
  Hierarchical occurrence within efficacy assessment time interval (EATI) of:
Change in KCCQ relative to baseline | 12 months
  Hierarchical occurrence within efficacy assessment time interval (EATI) of:

SECONDARY OUTCOMES:
MACCE defined as the composite of all-cause death, all stroke, and hospitalizations for heart failure or symptomatic aortic valve disease or clinically significant worsening of heart failure within EATI. Hierarchical occurrence within EATI of: | 12 month
  1. All-cause death
  2. Disabling stroke
  3. Hospitalizations related to heart failure, symptomatic aortic valve disease or non-disabling stroke or clinically significant worsening of heart failure (heart failure event)
-All-cause death within EATI | 12 month
  -All-cause death within EATI

CONTACTS AND LOCATIONS:
Locations (51):
- United States (46):
  - Chandler Regional Medical Center, Chandler, Arizona
  - UCSD/Sulpizio Cardiovascular Center, La Jolla, California
  - University of Southern California - Los Angeles, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - St. Joseph Hospital, Orange, California
  - UCSF, San Francisco, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Yale University, New Haven, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Advocate Christ Hospital, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Evanston Hospital/NorthShore Univ. Health System, Evanston, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Maine Medical Center, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beaumont Hospital, Royal Oak, Michigan
  - Ascension St. Mary's Hospital, Saginaw, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - HealthEast Medical Research Institute, Saint Paul, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morristown Memorial, Morristown, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Oregon Health Science University (OHSU), Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - PinnacleHealth Cardiovascular Institute, Wormleysburg, Pennsylvania
  - WellSpan York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt Heart and Vascular, Nashville, Tennessee
  - Seton Medical Center Austin, Austin, Texas
  - IHC Health Services, Inc. dba Intermountain Medical Center, Murray, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University (VCU), Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Oklahoma Heart Hospital, Milwaukee, Wisconsin
  - Advocate Aurora- St. Lukes, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- St. Michael's Hospital, Toronto, Ontario, Canada
- Netherlands (4):
  - University Medical Center Utrecht, Utrecht, TH
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam
  - Isala Clinics, Zwolle

REFERENCES:
- [Derived] Esquitin KA, Khalique OK, Liu Q, Kodali SK, Marcoff L, Nazif TM, George I, Vahl TP, Leon MB, Hahn RT. Accuracy of the Single Cycle Length Method for Calculation of Aortic Effective Orifice Area in Irregular Heart Rhythms. J Am Soc Echocardiogr. 2019 Mar;32(3):344-350. doi: 10.1016/j.echo.2018.11.018. Epub 2019 Jan 28. PMID 30704832